CLINICAL TRIAL: NCT00973128
Title: Reduced Doses of Antimony Plus Recombinant Human GM-CSF Compared With Antimony in Standard Doses for Cutaneous Leishmaniasis: a Randomized, Single-blind, Placebo-controlled, Pilot Study
Brief Title: Reduced Doses of Antimony Plus Ranulocyte Monocyte Colony Stimulating Factor (GM-CSF) for Cutaneous Leishmaniasis
Acronym: GMCSFSbv
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado da Bahia (Other)
Responsible Party: Roque Pacheco de Almeida, Hospital Universitário Prof. Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMCSFAntimonyCL
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — sargramostim; Meglumine Antimoniate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1: Cutaneous leishmaniasis patients randomized in Corte to receive antimony (20mg/daily for 10 days) plus GM-CSF Treatment: antimony (20mg/daily for 10 days) plus GM-CSF (400 µg, divided in two doses a week apart)
  Interventions: Drug: GMCSF plus Antimony reduced dose
- Group 2 (Active Comparator): Group 2: antimony in standard dose plus saline administered in an identical fashion to the GM-CSF.
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: GMCSF plus Antimony reduced dose — 400 µg, divided in two doses a week apart, antimony (20mg/daily for 10 days)
  Other Names: Sargramostim
  Arms: Group 1
Drug: Meglumine antimoniate — 20mg/daily for 20 days
  Other Names: pentavalent antimony
  Arms: Group 2

SUMMARY:
The present study was designed as a randomized, single blind, placebo-controlled, study to evaluate the effect of 400 µg of recombinant human GM-CSF applied intralesionally and associated with half of the total dose of antimony in a reduced time schedule (20mgSbV/Kg/d for 10 days) as compared to the full dose of antimony (20mgSbV/Kg/d for 20 days) to treat cutaneous leishmaniasis ulcers.

DETAILED DESCRIPTION:
This is a randomized, single blind placebo-controlled study in which the groups were selected from the cases presenting to the health post. The inclusion criteria were: age between 15 and 50 years, of either sex, diagnosis of cutaneous leishmaniasis of less than 60 days. The diagnostic criteria were the presence of a typical single cutaneous ulcer, localized on lower limbs, and a positive delayed type hypersensitivity test (DTH or Montenegro skin test) to Leishmania antigen.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 50 years
* Either gender
* Diagnosis of cutaneous leishmaniasis
* Less than 60 days of disease

Exclusion Criteria:

* Any history of prior anti-leishmania therapy
* Negative parasitology (aspirate/smear)or negative Montenegro test
* Pregnancy
* Age below 15 and above 50 years
* Other associated acute or chronic illnesses
* History of allergy to GM-CSF and/or antimony
* HIV, HTLV-1 infections or diabetes
* Administrative reasons:
* Lack of ability or willingness to give informed consent (patient and/or parent / legal representative)
* Anticipated non-availability for study visits/procedures

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2004-02; Primary Completion 2006-10 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Cure rate or complete cicatrization of the ulcer | 3 months after treatment

SECONDARY OUTCOMES:
Initial cure rate or complete cicatrization of the ulcer. | 2 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Roque P Almeida, MD, PhD, Principal Investigator — Hospital Universitário Prof Edgard Santos-UFBA
Locations (1):
- Health Post of Corte de Pedra, Valença, Estado de Bahia, Brazil